CLINICAL TRIAL: NCT01698619
Title: Hemodynamic Changes in Altitude Adaptation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Peter Stein, Consultant, Goethe University
Other Study IDs: AconcaguaIron
Record Dates: First submitted 2012-09-27; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Acute Mountain Sickness; High Altitude Pulmonary Edema; High Altitude Cerebral Edema
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Climbers on Mount Aconcagua: The Cohort consists of volunteers climbing Mount Aconcagua.

SUMMARY:
We use a new technology (Nexfin from BMEYE-Inventive Hemodynamics) to monitor Cardiac Output, Blood Pressure, Fluid Responsiveness, Pulse Oximetry, Hemoglobin Concentration, Oxygen Delivery in Climbers during their process of acclimatization on a expedition to Mount Aconcagua.

DETAILED DESCRIPTION:
Several parameters will be recorded to analyze their influence on the adaptation to high altitude. Such as, food composition, dietary supplements, water intake and output.

ELIGIBILITY:
Inclusion Criteria:

* No acute or chronic disease
* Body mass index : 20 - 30

Exclusion Criteria:

* Any preexisting disease that has a potential impact on physical performance such as:

  * pulmonary
  * cerebral
  * muscular
  * cardiac
  * vascular - diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers taking part in an expedition to Mount Aconcagua
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in Oxygen Delivery | daily, up to 18 days
  Unit: ml/min baseline measure will be obtained at sea level

SECONDARY OUTCOMES:
Changes from baseline in Hemoglobin Concentration | daily, up to 18 days
  Unit: mg/dl baseline measure will be obtained at sea level

OTHER OUTCOMES:
Changes from baseline in Blood pressure, Fluid Responsiveness, Oxygen Saturation, Cardiac Output | daily, up to 18 days
  baseline measure will be obtained at sea level

CONTACTS AND LOCATIONS:
Locations (1):
- Goethe University, Frankfurt am Main, Hesse, Germany